CLINICAL TRIAL: NCT02883556
Title: Phase II Study of Pembrolizumab (MK-3475) as First Line Single Drug Therapy in Patients With Unresectable Squamous Cell Carcinoma of the Skin
Brief Title: Study of Pembrolizumab as First Line Therapy in Patients With Unresectable Squamous Cell Carcinoma of the Skin
Acronym: CARSKIN
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P151202; 2016-002076-28 (EudraCT Number)
Record Dates: First submitted 2016-08-25; First posted 2016-08-30 (Estimated); Last update posted 2021-01-13 (Actual); Status verified 2020-07

CONDITIONS: Carcinoma, Squamous Cell
Keywords: Carcinoma; Squamous Cell; Skin; pembrolizumab; Programmed Cell Death 1 Ligand 1
MeSH Terms: conditions — Carcinoma, Squamous Cell; Carcinoma | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pembrolizumab 200 mg (Experimental): Pembrolizumab 200 mg administered as intravenous (IV) infusion every 3 weeks up to 24 months or until progression or unacceptable toxicity develops.
  Interventions: Drug: Pembrolizumab

INTERVENTIONS:
Drug: Pembrolizumab — 200 mg, administered as intravenous (IV) infusion every 3 weeks up to 24 months or until progression or unacceptable toxicity develops.
  Other Names: MK-3475, KEYTRUDA

SUMMARY:
The purpose of this study is to assess the efficacy and safety of pembrolizumab in patient with locally advanced or metastatic squamous cell carcinoma of the skin

DETAILED DESCRIPTION:
Agents blocking the Programmed Cell Death 1(PD1)/Programmed Cell Death 1-Ligand 1 (PD-L1) pathway have demonstrated objective, durable tumor regressions in patients with advanced solid malignancies and efficacy has been linked to PD-L1 expression. PD-L1 expression by tumour cells is the strongest single predictor of response to anti-PD1 therapy (J Taube, R Anders et al, Clin Cancer Res 2014). Pembrolizumab (MK-3475) is a high-affinity humanized monoclonal anti-PD1 antibody. It leads to dual PD1-ligand blockade of PD-L1 and PD-L2 that may reactivate the immune surveillance and elicit anti-tumour response. It has antitumor activity in melanoma and NSCLC (phase III trials). Pembrolizumab might be of interest in unresectable squamous cell carcinomas of the skin (SCCS).

Approximately 20% to 30% of non-melanoma skin cancers are SCCS. Most patients with primary SCCS have an excellent prognosis, but SCCS can progress to advanced stages that are impossible to treat by surgical excision or radiotherapy. Few therapeutic options are available for these tumors. Conventional chemotherapy, such as cisplatin-based combinations, has some efficacy, but the toxic effects of these combinations often prohibit their use in elderly patients. Epidermal Growth Factor (EGFR) signaling antagonists have activity only in a subset of patients. New therapeutic options are needed for patients with advanced SCCS.

No trial evaluating pembrolizumab in human SCCS is ongoing. Investigators hypothesize that:

i) PD-L1 is expressed in SCCS as in HNSCC ii) pembrolizumab may be effective as a single agent in patients with unresectable SCCS iii) Efficacy of pembrolizumab is correlated to PD-L1 expression in SCCS.

Investigators therefore intend to determine the efficacy and safety of single agent pembrolizumab in all patients and in patients with PD-L1-positive unresectable SCCS naïve of chemotherapy and of EGFR inhibitors.

ELIGIBILITY:
Inclusion Criteria:

* Be willing and able to provide written informed consent/assent for the trial
* Be more than 18 years of age on day of signing informed consent.
* Be either affiliated to, or a beneficiary of, a social security category
* Have metastatic disease, or locally advanced disease not amenable to surgery with documented progression
* Be willing and able to undergo pre-treatment baseline biopsy of the tumor
* PD-L1+ or PD-L1- tumors
* Have measurable disease based on RECIST 1.1
* Have a performance status of 0 or 1 on the Easter Cooperative Oncology Group (ECOG) Performance Scale.
* Demonstrate adequate organ function as defined in Table 3, all screening labs should be performed within 10 days of treatment initiation.
* Have recovered from major surgery or radiation therapy
* Female subject of childbearing potential should have a negative urine or serum pregnancy test within 72 hours prior to receiving the first dose of study medication.
* Female subjects of childbearing potential should be willing to use 1 method of birth control before the first dose of study therapy through 120 days after the last dose of study therapy. (Reference Section 7.5.1).

Male subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy.

Exclusion Criteria:

* Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks or 5 half-lives (minimum 14 days), whichever is shorter, prior to the first dose of treatment.
* Has received prior therapy with either chemotherapy or targeted therapy for the present tumor
* Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent.
* Has received radiation therapy within 4 weeks prior to study Day 1
* Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
* Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies)
* Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., Hepatitis C Virus RNA [qualitative] is detected).
* Has known history of, or any evidence of active, non-infectious pneumonitis.
* Has an active infection requiring systemic therapy
* Has received a live vaccine within 30 days of planned start of study therapy.
* Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Fluenz tetra®) are live attenuated vaccines, and are not allowed.
* Hypersensitivity to pembrolizumab or any of its excipients.
* Has a known additional malignancy. Exceptions include i) basal cell carcinoma of the skin or other squamous cell carcinoma of the skin or in situ cervical cancer, ii) history of another non blood malignancy that has undergone potentially curative therapy without recurrence for more than 2 years.
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with brain metastases may participate provided they are stable (without evidence of progression by imaging for at least eight weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment. This exception does not include carcinomatous meningitis which is excluded regardless of clinical stability.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2017-03-27 (Actual); Primary Completion 2019-03-23 (Actual); Study Completion 2020-12-15 (Actual)

PRIMARY OUTCOMES:
Response rate (RR) | 15 weeks
  Response rate (RR) at 15 weeks (RECIST v.1.1) in the whole sample by CT or MRI Response Evaluation Criteria in Solid Tumors with central radiology review

SECONDARY OUTCOMES:
Safety profile (NCI CTCAE v4.0) | up to 28 months
  Advers event and serious adverse event status
RR in PD-L1-positive patients | 15 weeks
  To assess in the whole sample and in PD-L1 positive patients
Disease Control Rate using RECIST and modified RECIST v.1.1 | 15 weeks
  Controled by the radiological evaluation
RR using modified RECIST 1.1 | 15 weeks
  Controled by the radiological evaluation
RR using RECIST and modified RECIST v.1.1 | 24 weeks
  Controled by the radiological evaluation
Best RR using RECIST and modified RECIST v.1.1 | 24 months
  The best response was collected after all radiological evaluation completion
Overall Survival (OS) | up to 24 months
  Survival status
Progression Free Survival by RECIST 1.1 and modified RECIST 1.1 | up to 24 months
  Controled by the radiological evaluation
Duration of response (DOR) by RECIST 1.1 and modified RECIST 1.1 | up to 24 months
  Controled by the radiological evaluation
Duration of control by RECIST 1.1 and modified RECIST 1.1 | up to 24 months
  Controled by the radiological evaluation
Time to disease progression by RECIST 1.1 and modified RECIST 1.1 | up to 24 months
  Controled by the radiological evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Eve MAUBEC, Pr, Principal Investigator — Assistance Publique - Hôpitaux de Paris; Zahia Ben-Abdesselam, CP, Study Director — Unité de Recherche clinique
Locations (1):
- Hôpital Avicenne, Bobigny, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Maubec E, Boubaya M, Petrow P, Beylot-Barry M, Basset-Seguin N, Deschamps L, Grob JJ, Dreno B, Scheer-Senyarich I, Bloch-Queyrat C, Leccia MT, Stefan A, Saiag P, Grange F, Meyer N, de Quatrebarbes J, Dinulescu M, Legoupil D, Machet L, Dereure O, Zehou O, Montaudie H, Wierzbicka-Hainaut E, Le Corre Y, Mansard S, Guegan S, Arnault JP, Dalac S, Aubin F, Alloux C, Lopez I, Cherbal S, Tibi A, Levy V; Groupe de Cancerologie Cutanee30. Phase II Study of Pembrolizumab As First-Line, Single-Drug Therapy for Patients With Unresectable Cutaneous Squamous Cell Carcinomas. J Clin Oncol. 2020 Sep 10;38(26):3051-3061. doi: 10.1200/JCO.19.03357. Epub 2020 Jul 30. PMID 32730186